CLINICAL TRIAL: NCT05001438
Title: Aleatorized Prospective Study on the Eficacy of Movilization Under Anesthesia in Patients With Frozen Shoulder That Already Receive Treatment With Hidrodilatation.
Brief Title: MUA's Efficacy in Frozen Shoulder in Patients Which Already Received an Hidrodilatation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2021/0567
Record Dates: First submitted 2021-07-19; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hidro alone (Active Comparator): The patient receives the Hidrodilatation guided by ultrasonography under anesthetic blockage of the circumflex nerve and the supraescapular nerve. The hidrodilatation is achieved by insuflating the articulation with 2 cc of trigon depot + 10 cc 1% mepivacain + 11 cc saline serum.
  Interventions: Procedure: Hidro
- Hidro + MUA (Experimental): The patient receives the Hidrodilatation guided by ultrasonography under anesthetic blockage of the circumflex nerve and the supraescapular nerve. The hidrodilatation is achieved by insuflating the articulation with 2 cc of trigon depot + 10 cc 1% mepivacain + 11 cc saline serum.
  After the Hidrodilatation the patient is sedated and then a Movilization of the glenohumeral joint is performed.
  Interventions: Procedure: Hidro; Procedure: MUA

INTERVENTIONS:
Procedure: Hidro — Guided by ultrasonography under anesthetic blockage of the circumflex nerve and the supraescapular nerve. The hidrodilatation is achieved by insuflating the articulation with 2 cc of trigon depot + 10 cc 1% mepivacain + 11 cc saline serum.
Procedure: MUA — Movilization under anesthesia
  Arms: Hidro + MUA

SUMMARY:
Hidrodilatation alone is as efective as Hidrodilatation + Movilization under anesthesia to treat the frozen shoulder

DETAILED DESCRIPTION:
"Frozen shoulder" disease is a pathological entity defined by the presence of a painful shoulder accompanied by restricted mobility. It affects 2% of the population with a slight predominance in women and the average age ranges between 40 and 60 years. The diagnosis of frozen shoulder is clinical and by exclusion; it presents with constant pain, especially at night, which increases on sudden mobilization, with restriction of at least two axes of shoulder mobility, especially external rotation and abduction.

The initial treatment of these patients is always conservative and consists of the association of pharmacological treatment (analgesics and anti-inflammatory drugs) together with a specific rehabilitation program. However, in many cases recovery is not complete and many patients require additional more invasive treatments.

Hydrodilation is a technique described in 1965 that consists of infiltrating 20-40 cc of serum into the glenohumeral joint to distend the joint capsule. In most cases, it is also associated with intra-articular corticosteroid and anesthetic infiltration to add an anti-inflammatory and anesthetic effect to joint distention. Several studies have shown good results with this treatment, however, many patients persist with pain and significant functional limitations despite this treatment.

Joint Mobilization Under general Anesthesia (MUA) is a more invasive alternative therapeutic technique that consists of a controlled mobilization under general anesthesia to break the synovial adhesions and the joint capsule, with the objective of increasing the range of motion. Several studies have evaluated the effectiveness and safety of this treatment, considered today a valid option for the treatment of frozen shoulder refractory to more conservative treatment.

Some studies have already compared the effectiveness of hydrodilatation with MUA as treatments for frozen shoulder. Jacob et al. demonstrated the same effectiveness between hydrodilatation and MUA, however, MUA reported a higher rate of iatrogenesis: hemarthrosis and lesions in the labrum, glenohumeral ligament or subscapularis ligament. However, there is no study evaluating the synergy of both techniques in the treatment of painful shoulder.

The aim of the present study is to assess the clinical efficacy of the combination of hydrodilatation and MUA in patients with frozen shoulder and to compare it with hydrodilatation alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient with "frozen shoulder", defined as painful shoulder accompanied with a greater or lesser degree of restriction of mobility, especially in passive external rotation of at least 3 months of evolution. The diagnosis, according to the usual protocol of the unit, should include radiological images that rule out degenerative or necrotic pathology and the performance of an ultrasound or MRI to rule out associated pathology of the rotator cuff, which are already obtained in the usual clinical follow-up.
* Failure of conservative treatment after a period of 3 months.
* Acceptance and signature of informed consent.

Exclusion Criteria:

* Known allergies to corticosteroids
* Patients with frozen shoulder secondary to previous shoulder surgery.
* High-risk patients in need of anticoagulant treatments.
* Patients with previous shoulder fracture.
* History of joint infection.
* Active neoplastic process.
* Associated rheumatic pathology.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Dissability Index | 1 year
  13 items completed by the patient on shoulder pain and function. A score of 0 indicates best 100 indicates worst

CONTACTS AND LOCATIONS:
Overall Officials: GUILLEM CLARET, PhD, Principal Investigator — Specialty surgeon
Locations (1):
- Hospital Clínic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The intention is to publish the study findings in an international journal of the specialty.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Publication by 2023
Access Criteria: Open access vs private peer reviewed journal